CLINICAL TRIAL: NCT03885596
Title: An Open-Label Study of Intraoperative CA-008 Administration in Subjects Undergoing Bunionectomy
Brief Title: Open-Label CA-008 (Vocacapsaicin) in Bunionectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Concentric Analgesics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA-PS-205
Record Dates: First submitted 2019-03-20; First posted 2019-03-21 (Actual); Results first posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Ketorolac; Fentanyl; Bupivacaine; Lidocaine; Celecoxib; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CA-008 Cohort 1 (Experimental): CA-008 4.2 mg reconstituted in saline
  All subjects received monitored anesthesia care (MAC) and a Mayo block followed by a sciatic (popliteal) nerve block.
  Interventions: Drug: CA-008; Drug: Ketorolac; Drug: Acetaminophen IV; Drug: Fentanyl; Drug: Bupivacaine Hydrochloride; Drug: Lidocaine HCl; Drug: Celecoxib; Drug: Acetaminophen Oral
- CA-008 Cohort 2 (Experimental): CA-008 4.2 mg reconstituted in saline
  All subjects received monitored anesthesia care (MAC) and a Mayo block.
  Interventions: Drug: CA-008; Drug: Ketorolac; Drug: Acetaminophen IV; Drug: Fentanyl; Drug: Bupivacaine Hydrochloride; Drug: Celecoxib; Drug: Acetaminophen Oral; Drug: Lidocaine Hydrochloride
- CA-008 Cohort 3 (Experimental): CA-008 4.2 mg reconstituted in saline
  All subjects received monitored anesthesia care (MAC) and a Mayo block.
  Interventions: Drug: CA-008; Drug: Ketorolac; Drug: Acetaminophen IV; Drug: Fentanyl; Drug: Bupivacaine Hydrochloride; Drug: Lidocaine Hydrochloride
- Exparel (Active Comparator): 106 mg [8 mL of the 133 mg/10 mL suspension] only
  All subjects received monitored anesthesia care (MAC) and a Mayo block.
  Interventions: Drug: Ketorolac; Drug: Acetaminophen IV; Drug: Fentanyl; Drug: Bupivacaine Hydrochloride; Drug: Lidocaine Hydrochloride; Drug: Exparel

INTERVENTIONS:
Drug: CA-008 — Drug: CA-008 4.2 mg reconstituted in saline
  Other Names: Vocacapsaicin
  Arms: CA-008 Cohort 1; CA-008 Cohort 2; CA-008 Cohort 3
Drug: Ketorolac — 30 mg IV at the onset of anesthesia
Drug: Acetaminophen IV — 1 g at the onset of anesthesia
Drug: Fentanyl — 100 mcg IV fentanyl administered at the onset of anesthesia and additional 50 mcg near the end of surgery
Drug: Bupivacaine Hydrochloride — 0.25% 30 mL (75 mg) prior to surgery
Drug: Lidocaine HCl — 1.5% 12 mL at the end of surgery
  Arms: CA-008 Cohort 1
Drug: Celecoxib — 200 mg PO bid each day postoperative
  Arms: CA-008 Cohort 1; CA-008 Cohort 2
Drug: Acetaminophen Oral — 1 g postoperative
  Arms: CA-008 Cohort 1; CA-008 Cohort 2
Drug: Lidocaine Hydrochloride — 2% 15 mL at the end of surgery
  Arms: CA-008 Cohort 2; CA-008 Cohort 3; Exparel
Drug: Exparel — Bupivacaine liposome injection suspension
  Arms: Exparel

SUMMARY:
A Phase 2, open-label study of CA-008 to evaluate post-surgical pain control with CA-008.

DETAILED DESCRIPTION:
This is a Phase 2, single-center, open-label study evaluating a single dose of CA-008 4.2 mg administered with different standard-of-care anesthetic regimens during an elective unilateral transpositional first metatarsal osteotomy for the correction of hallux valgus deformity (bunionectomy).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult aged 18 - 65 years old
2. American Society of Anesthesiology (ASA) physical Class 1, 2 or 3
3. Planning elective Bunionectomy repair
4. For both males and females: using an acceptable method of birth control
5. If a female: not pregnant or breastfeeding
6. Have a body mass index ≤ 36 kg/m2

Exclusion Criteria:

1. Have another painful condition, other than bunion-related pain, that may require pain treatment during the study period
2. Have active skin disease or another abnormality at the anticipated site of surgery that could interfere with the planned surgery.
3. Have a known allergy to study medications.
4. Have a history of significant medical, neuropsychiatric or other condition, including a clinically significant abnormal clinical laboratory test values
5. Have positive results on the alcohol test (breath or saliva) or urine drug screen.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Wu, Study Director — Concentric Analgesics
Locations (1):
- Lotus Clinical Research, LLC, Pasadena, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- CA-008 Cohort 1: CA-008 4.2 mg
  All subjects received monitored anesthesia care (MAC) and a Mayo block followed by a sciatic (popliteal) nerve block.
  CA-008: Drug: CA-008 4.2 mg
  Ketorolac: 30 mg IV at the onset of anesthesia
  Acetaminophen IV: 1 g at the onset of anesthesia
  Fentanyl: 100 mcg IV fentanyl administered at the onset of anesthesia and additional 50 mcg near the end of surgery
  Bupivacaine Hydrochloride: 0.25% 30 mL (75 mg) prior to surgery
  Lidocaine HCl: 1.5% 12 mL at the end of surgery
  Celecoxib: 200 mg PO bid each day postoperative
  Acetaminophen Oral: 1 g postoperative
- CA-008 Cohort 2: CA-008 4.2 mg
  All subjects received monitored anesthesia care (MAC) and a Mayo block.
  CA-008: Drug: CA-008 4.2 mg
  Ketorolac: 30 mg IV at the onset of anesthesia
  Acetaminophen IV: 1 g at the onset of anesthesia
  Fentanyl: 100 mcg IV fentanyl administered at the onset of anesthesia and additional 50 mcg near the end of surgery
  Bupivacaine Hydrochloride: 0.25% 30 mL (75 mg) prior to surgery
  Celecoxib: 200 mg PO bid each day postoperative
  Acetaminophen Oral: 1 g postoperative
  Lidocaine Hydrochloride: 2% 15 mL at the end of surgery
- CA-008 Cohort 3: CA-008 4.2 mg
  All subjects received monitored anesthesia care (MAC) and a Mayo block.
  CA-008: Drug: CA-008 4.2 mg
  Ketorolac: 30 mg IV at the onset of anesthesia
  Acetaminophen IV: 1 g at the onset of anesthesia
  Fentanyl: 100 mcg IV fentanyl administered at the onset of anesthesia and additional 50 mcg near the end of surgery
  Bupivacaine Hydrochloride: 0.25% 30 mL (75 mg) prior to surgery
  Lidocaine Hydrochloride: 2% 15 mL at the end of surgery
- Exparel: 106 mg [8 mL of the 133 mg/10 mL suspension] only
  All subjects received monitored anesthesia care (MAC) and a Mayo block.
  Ketorolac: 30 mg IV at the onset of anesthesia
  Acetaminophen IV: 1 g at the onset of anesthesia
  Fentanyl: 100 mcg IV fentanyl administered at the onset of anesthesia and additional 50 mcg near the end of surgery
  Bupivacaine Hydrochloride: 0.25% 30 mL (75 mg) prior to surgery
  Lidocaine Hydrochloride: 2% 15 mL at the end of surgery
  Exparel: Bupivacaine liposome injection suspension
Period: Overall Study
Arm/Group | CA-008 Cohort 1 | CA-008 Cohort 2 | CA-008 Cohort 3 | Exparel
Started | 9 | 9 | 9 | 9
Completed | 7 | 8 | 9 | 9
Not Completed | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- CA-008 (Vocacapsaicin) Cohort 1: CA-008 4.2 mg reconstituted in saline
  All subjects received monitored anesthesia care (MAC) and a Mayo block followed by a sciatic (popliteal) nerve block.
  CA-008: Drug: CA-008 4.2 mg reconstituted in saline
  Ketorolac: 30 mg IV at the onset of anesthesia
  Acetaminophen IV: 1 g at the onset of anesthesia
  Fentanyl: 100 mcg IV fentanyl administered at the onset of anesthesia and additional 50 mcg near the end of surgery
  Bupivacaine Hydrochloride: 0.25% 30 mL (75 mg) prior to surgery
  Lidocaine HCl: 1.5% 12 mL at the end of surgery
  Celecoxib: 200 mg PO bid each day postoperative
  Acetaminophen Oral: 1 g postoperative
- CA-008 (Vocacapsaicin) Cohort 2: CA-008 4.2 mg reconstituted in saline
  All subjects received monitored anesthesia care (MAC) and a Mayo block.
  CA-008: Drug: CA-008 4.2 mg reconstituted in saline
  Ketorolac: 30 mg IV at the onset of anesthesia
  Acetaminophen IV: 1 g at the onset of anesthesia
  Fentanyl: 100 mcg IV fentanyl administered at the onset of anesthesia and additional 50 mcg near the end of surgery
  Bupivacaine Hydrochloride: 0.25% 30 mL (75 mg) prior to surgery
  Celecoxib: 200 mg PO bid each day postoperative
  Acetaminophen Oral: 1 g postoperative
  Lidocaine Hydrochloride: 2% 15 mL at the end of surgery
- CA-008 (Vocacapsaicin) Cohort 3: CA-008 4.2 mg reconstituted in saline
  All subjects received monitored anesthesia care (MAC) and a Mayo block.
  CA-008: Drug: CA-008 4.2 mg reconstituted in saline
  Ketorolac: 30 mg IV at the onset of anesthesia
  Acetaminophen IV: 1 g at the onset of anesthesia
  Fentanyl: 100 mcg IV fentanyl administered at the onset of anesthesia and additional 50 mcg near the end of surgery
  Bupivacaine Hydrochloride: 0.25% 30 mL (75 mg) prior to surgery
  Lidocaine Hydrochloride: 2% 15 mL at the end of surgery
- Total: Total of all reporting groups
Arm/Group | CA-008 (Vocacapsaicin) Cohort 1 | CA-008 (Vocacapsaicin) Cohort 2 | CA-008 (Vocacapsaicin) Cohort 3 | Exparel | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (9.96) | 43.1 (9.20) | 35.2 (12.71) | 52.8 (6.72) | 45.05 (9.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 8 | 5 | 27
  Male | 2 | 2 | 1 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6 | 4 | 16
  Not Hispanic or Latino | 5 | 7 | 3 | 5 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 2 | 4 | 2 | 2 | 10
  White | 6 | 4 | 6 | 7 | 23
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 9 | 9 | 36

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of Numerical Rating Scale (NRS) Scores (at Rest) Over 72h
Description: Area Under the Curve of pain intensity scores (using a Numeric Rating Scale of pain intensity from 0-10 where 0 is no pain and 10 is the worst pain imaginable) over 72 hours
Time Frame: 0-72 hours
Population: Safety population
Measure: Mean (Standard Deviation); unit: score on a scale*hour
Groups:
- CA-008 Cohort 1: CA-008 4.2 mg reconstituted in saline
  All subjects received monitored anesthesia care (MAC) and a Mayo block followed by a sciatic (popliteal) nerve block.
  CA-008: Drug: CA-008 4.2 mg reconstituted in saline
  Ketorolac: 30 mg IV at the onset of anesthesia
  Acetaminophen IV: 1 g at the onset of anesthesia
  Fentanyl: 100 mcg IV fentanyl administered at the onset of anesthesia and additional 50 mcg near the end of surgery
  Bupivacaine Hydrochloride: 0.25% 30 mL (75 mg) prior to surgery
  Lidocaine HCl: 1.5% 12 mL at the end of surgery
  Celecoxib: 200 mg PO bid each day postoperative
  Acetaminophen Oral: 1 g postoperative
- CA-008 Cohort 2: CA-008 4.2 mg reconstituted in saline
  All subjects received monitored anesthesia care (MAC) and a Mayo block.
  CA-008: Drug: CA-008 4.2 mg reconstituted in saline
  Ketorolac: 30 mg IV at the onset of anesthesia
  Acetaminophen IV: 1 g at the onset of anesthesia
  Fentanyl: 100 mcg IV fentanyl administered at the onset of anesthesia and additional 50 mcg near the end of surgery
  Bupivacaine Hydrochloride: 0.25% 30 mL (75 mg) prior to surgery
  Celecoxib: 200 mg PO bid each day postoperative
  Acetaminophen Oral: 1 g postoperative
  Lidocaine Hydrochloride: 2% 15 mL at the end of surgery
- CA-008 Cohort 3: CA-008 4.2 mg reconstituted in saline
  All subjects received monitored anesthesia care (MAC) and a Mayo block.
  CA-008: Drug: CA-008 4.2 mg reconstituted in saline
  Ketorolac: 30 mg IV at the onset of anesthesia
  Acetaminophen IV: 1 g at the onset of anesthesia
  Fentanyl: 100 mcg IV fentanyl administered at the onset of anesthesia and additional 50 mcg near the end of surgery
  Bupivacaine Hydrochloride: 0.25% 30 mL (75 mg) prior to surgery
  Lidocaine Hydrochloride: 2% 15 mL at the end of surgery
Arm/Group | CA-008 Cohort 1 | CA-008 Cohort 2 | CA-008 Cohort 3 | Exparel
Number analyzed (Participants) | 9 | 9 | 9 | 9
score on a scale*hour | 72.30 (95.476) | 66.24 (54.365) | 203.76 (103.718) | 306.58 (92.883)

2. Secondary Outcome: Opioid Consumption
Description: Summary of opioid consumption in oral morphine equivalents
Time Frame: 0-72 hours
Population: Safety population
Measure: Mean (Standard Deviation); unit: mg morphine equivalents
Arm/Group | CA-008 (Vocacapsaicin) Cohort 1 | CA-008 (Vocacapsaicin) Cohort 2 | CA-008 (Vocacapsaicin) Cohort 3 | Exparel
Number analyzed (Participants) | 9 | 9 | 9 | 9
mg morphine equivalents | 10.83 (27.33) | 3.33 (6.61) | 38.33 (26.90) | 80.83 (66.95)

3. Primary Outcome: Pain Intensity Scores at 24 Hours at Rest Using Numerical Rating Scale (NRS)
Description: Numeric Rating Scale (NRS) of pain intensity from 0-10 where 0 is no pain and 10 is the worst pain imaginable at 24 hours
Time Frame: 24 hours
Population: Safety population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CA-008 Cohort 1 | CA-008 Cohort 2 | CA-008 Cohort 3 | Exparel
Number analyzed (Participants) | 9 | 9 | 9 | 9
units on a scale | 0.6 (0.88) | 1.7 (1.66) | 5.1 (1.45) | 6.0 (1.00)

4. Primary Outcome: Pain Intensity Scores at 48 Hours at Rest Using Numerical Rating Scale (NRS)
Description: Numeric Rating Scale (NRS) of pain intensity from 0-10 where 0 is no pain and 10 is the worst pain imaginable at 48 hours
Time Frame: 48 hours
Population: Safety population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CA-008 Cohort 1 | CA-008 Cohort 2 | CA-008 Cohort 3 | Exparel
Number analyzed (Participants) | 9 | 9 | 9 | 9
score on a scale | 1.3 (2.12) | 0.6 (0.73) | 2.7 (2.45) | 4.8 (2.11)

5. Primary Outcome: Pain Intensity Scores at 72 Hours at Rest Using Numerical Rating Scale (NRS)
Description: Numeric Rating Scale (NRS) of pain intensity from 0-10 where 0 is no pain and 10 is the worst pain imaginable at 72 hours
Time Frame: 72 hours
Population: Safety population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CA-008 Cohort 1 | CA-008 Cohort 2 | CA-008 Cohort 3 | Exparel
Number analyzed (Participants) | 9 | 9 | 9 | 9
score on a scale | 1.2 (2.28) | 0.3 (0.71) | 2.0 (2.12) | 4.6 (2.88)

ADVERSE EVENTS:
Time Frame: Up to 76 days: Screening period from 45 days prior to surgery (D-45) to D29±2 Study Completion Visit. Unscheduled visits or visits after D29 might be necessary to assess ongoing safety issues or to follow an event to resolution or to establishment of a new baseline.
Arm/Group | CA-008 Cohort 1 | CA-008 Cohort 2 | CA-008 Cohort 3 | Exparel
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 1/9 | 4/9 | 5/9 | 5/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CA-008 Cohort 1 (N=9) | CA-008 Cohort 2 (N=9) | CA-008 Cohort 3 (N=9) | Exparel (N=9)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Sensory disturbance (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT03885596/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/96/NCT03885596/SAP_001.pdf